CLINICAL TRIAL: NCT06371651
Title: Enhancing Brain Oxygenation: Effects of Short-Term Co-Administration of Creatine and Guanidinoacetic Acid at Rest and During Stress
Brief Title: Creatine and GAA for Brain Oxygenation
Acronym: CREGAA-OXY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Professor, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 23-1462-3
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Oxygen Deficiency
Keywords: creatine; guanidinoacetic acid; oxygen saturation; brain
MeSH Terms: conditions — Hypoxia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Experimental): One sachet of supplement before breakfast and dinner
  Interventions: Dietary Supplement: Supplement
- Placebo (Placebo Comparator): One sachet of inert compound before breakfast and dinner
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement — Dietary supplement containing creatine and guanidinoacetic acid
  Arms: Supplement
Dietary Supplement: Placebo — Inert substance
  Arms: Placebo

SUMMARY:
The main aim of this randomized controlled trial is to evaluate cerebral blood oxygenation after 7-day administration of a creatine-guanidinoacetic acid (GAA) mixture in healthy adults before, during, and after a series of cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years
* Absence of metabolic disorders or other health complications
* Provision of signed informed consent

Exclusion Criteria:

* History of dietary supplement use within the preceding 4 weeks
* Lack of consent to randomization
* Concurrent participation in other studies

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Brain oxygen saturation | Change from baseline brain oxygen saturation at 2 weeks
  Percentage of oxygen saturation in prefrontal brain

SECONDARY OUTCOMES:
Hemoglobin index | Change from baseline hemoglobin index at 2 weeks
  Concentration of hemoglobin index in prefrontal brain

CONTACTS AND LOCATIONS:
Overall Officials: Sergej Ostojic, MD, PhD, Principal Investigator — University of Novi Sad
Locations (1):
- Applied Bioenergetics Lab at Faculty of Sport and PE, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in nutritional neuroscience. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be made accessible for up to 12 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Only qualified researchers with academic interest in in nutritional neuroscience

REFERENCES:
- [Background] Watanabe A, Kato N, Kato T. Effects of creatine on mental fatigue and cerebral hemoglobin oxygenation. Neurosci Res. 2002 Apr;42(4):279-85. doi: 10.1016/s0168-0102(02)00007-x. PMID 11985880
- [Background] Hammett ST, Wall MB, Edwards TC, Smith AT. Dietary supplementation of creatine monohydrate reduces the human fMRI BOLD signal. Neurosci Lett. 2010 Aug 2;479(3):201-5. doi: 10.1016/j.neulet.2010.05.054. Epub 2010 May 24. PMID 20570601
- [Derived] Zanini D, Todorovic N, Ostojic SM. Creatine with guanidinoacetic acid improves prefrontal brain oxygenation before, during, and after a cognitive task: A randomized controlled pilot trial. Nutr Health. 2025 Jun;31(2):363-368. doi: 10.1177/02601060241300236. Epub 2024 Nov 21. PMID 39569437
- See also: Web page of study lab — https://www.appliedbioenergetics.org/